CLINICAL TRIAL: NCT03602248
Title: Acute Effects of Two Different Speed Endurance Protocols on Performance, Muscle Damage Markers and Neuromuscular Fatigue in Soccer Players
Brief Title: Speed Endurance Training, Muscle Damage and Performance in Soccer Players
Acronym: SPENSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: SpEndu2018
Record Dates: First submitted 2018-06-12; First posted 2018-07-26 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Speed Endurance Training Protocol 1; Speed Endurance Training Protocol 2; Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Speed endurance training protocol A (Experimental): Performance of two different speed endurance training protocols:
  Speed endurance training protocol A will consist of 1 set of 8 repetitions interspersed by 2,5 minutes of recovery with a work to rest ratio of 1:5 (25-30 seconds all out work).
  Interventions: Other: Speed endurance training protocol A
- Speed endurance training protocol B (Experimental): Speed endurance training protocol B will consist of 1 set of 8 repetitions interspersed by 4 minutes of recovery with a work to rest ratio of 1:8 (25-30 seconds all out work)
  Interventions: Other: Speed endurance training protocol B
- Control condition (No Intervention): No training protocol will be performed, the participants will perform only the measurements for performance and muscle damage and neuromuscular fatigue

INTERVENTIONS:
Other: Speed endurance training protocol A — 1 set of 8 repetitions interspersed by 2,5 minutes of recovery with a work to rest ratio of 1:5 (25-30 seconds all out work)
  Arms: Speed endurance training protocol A
Other: Speed endurance training protocol B — 1 set of 8 repetitions interspersed by 4 minutes of recovery with a work to rest ratio of 1:8 (25-30 seconds all out work)
  Arms: Speed endurance training protocol B

SUMMARY:
Soccer is an intermittent sport in which the aerobic and anaerobic capacity of the players are both very important. Elite football players perform an average of 150-250 short and intense movements during a match, demonstrating the significant contribution of the anaerobic energy system. Speed endurance training consists a tool to enhance the performance of aerobic and anaerobic system. This training includes actions such as sprinting, changes of direction, accelerations, decelerations, jumps and shooting, characterized by a strong eccentric component. Eccentric actions are associated with exercise induced muscle damage (EIMD). Nevertheless, to date, EIMD responses following a session of speed endurance training have not yet been investigated. Therefore, the aim of the present study is to examine the EIMD responses and changes on performance and neuromuscular fatigue indices after two different speed endurance training protocols.

DETAILED DESCRIPTION:
Football is a team sport in which mean and maximum heart rate ranges from 85 to 98% of the maximum heart rate during a competitive match. Elite football players perform an average of 150-250 short and intense movements during a match while blood lactate values range from 2 to 14 mmol/L demonstrating that the anaerobic energy system contributes significantly during the game. Acceleration and deceleration ability as well as ability to perform repeated sprints and changes of direction greatly determine performance in soccer.

Soccer players' ability to perform repetitive high intensity sprints over a long period of time can be improved by speed endurance training. Speed endurance training consists of repetitive intense exercise bouts at a higher intensity than maximum aerobic speed (MAS) lasting from 10 to 40 seconds and has been proven to be an important tool for improving performance in trained soccer players. Improved performance is attributed to the muscle's increased regulatory capacity regarding intense exercise, enhanced recovery of the energy stores, increased activity and number of muscle enzymes and accelerated by-products removal, thereby contributing to the maintenance of homeostasis and delay of fatigue occurrence during intense exercise.

Speed endurance training includes repeated high intensity actions such as sprinting, changes of direction, accelerations, decelerations, jumps and shooting. However, these movements have a strong eccentric component which has been associated with exercise induced muscle damage (EIMD) and inflammation. EIMD increases plasma creatine kinase (CK) levels and the delayed onset of muscle soreness (DOMS) and reduces power production capacity. CK increases after a soccer match, peaks at 48 hours and returns to rest values 5-7 days after the match. DOMS increases immediately after a soccer match, peaks at 24-72 hours and is normalized ~5 days post match. The reduction in power production capacity is observed immediately after the match and remains reduced for ~72 hours with the largest decrease observed at 48 hours post-match. Nevertheless, to date, EIMD responses following a session of speed endurance training have not yet been investigated. Therefore, the aim of the proposed study is to examine the EIMD responses and changes on performance and neuromuscular fatigue indices after two speed endurance training protocols.

A preliminary power analysis (effect size >0.55, probability error of 0.05, power of 0.90) revealed that a total sample of 8-10 soccer players required to detect statistically meaningful differences after a speed endurance training protocol.

A randomized, three-trial (speed endurance protocol A vs. speed endurance protocol B vs. control), cross-over, repeated measures design will be implemented. The study will be performed one week after the end of the in-season to minimize the detraining effect. Prior to the first trial participants will have their body mass, height, body composition and performance measured and will be familiarized with all the testing procedures. Each experimental trial (speed endurance training protocol A and B) will include a speed endurance training session on Monday. The second trial (between training trials) will serve as control, where only performance measurements and blood sampling will be performed. Performance assessment and blood sampling will be performed immediately after each speed endurance training session and daily for three days post training session. Each training session will be performed on natural grass surface under the same environmental conditions (i.e. temperature and humidity). A 5-day recovery period will be used between trials. During the training sessions, participants will consume only water ad libitum. Field activity during training sessions will be recorded using high time-resolution Global Positioning System (GPS) instrumentation and heart rate monitoring. Before each training session, a standard breakfast and meal will be consumed by all players as previously described.

Speed endurance training protocols Speed endurance training protocol A will consist of 1 set of 8 repetitions interspersed by 2,5 minutes of recovery with a work to rest ratio of 1:5 (25-30 seconds all out work) whereas speed endurance training protocol B will consist of 1 set of 8 repetitions interspersed by 4 minutes of recovery with a work to rest ratio of 1:8 (25-30 seconds all out work). Both training protocols will include the same exercise (drill), consisting of multiple linear sprints, changes of direction, ball contacts, passes, and shooting. Prior to the training sessions, a 15-min standard warm-up (free running, active stretching, ball contacts and sprints) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any musculoskeletal injury for at least 6 months prior to the study
* No use of any drugs or ergogenic supplements for at least 6 months prior to the study
* Absence of regular soccer training for the last 3 years

Exclusion Criteria:

* Any recent incidence of musculoskeletal injury
* Use of any drugs or ergogenic supplements for the last 6 months
* Regular soccer training for the last 3 years

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Differences in changes in creatine kinase (CK) between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Creatine kinase (CK) is a muscle damage marker
Differences in changes in delayed onset of muscle soreness (DOMS) between the two training protocols | Pre-protocol, Day 1, Day 2, Day 3
  Delayed onset of muscle soreness (DOMS) is a muscle damage marker
Differences in changes in maximal concentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal concentric strength is used as a muscle damage marker
Differences in changes in maximal eccentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal eccentric strength is used as a muscle damage marker

SECONDARY OUTCOMES:
Differences in changes in countermovement jump between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Countermovement jump is used as a performance marker
Differences in changes in Repeated Sprint Ability (RSA) between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Repeated Sprint Ability (RSA) is a performance marker
Differences in changes in maximal concentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal concentric strength is used as a performance marker
Differences in changes in maximal eccentric strength between the two training protocols | Baseline, Day 1, Day 2, Day 3
  Maximal eccentric strength is used as a performance marker
Differences in changes in maximal isometric strength between the two training protocols | Baseline, Hour 1, Hour 2, Hour 3
  Maximal isometric strength is used as a neuromuscular fatigue marker

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Laboratory of Exercise Biochemistry, Exercise Physiology,and Sports Nutrition, School of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohr M, Krustrup P, Bangsbo J. Match performance of high-standard soccer players with special reference to development of fatigue. J Sports Sci. 2003 Jul;21(7):519-28. doi: 10.1080/0264041031000071182. PMID 12848386
- [Background] Ade JD, Harley JA, Bradley PS. Physiological response, time-motion characteristics, and reproducibility of various speed-endurance drills in elite youth soccer players: small-sided games versus generic running. Int J Sports Physiol Perform. 2014 May;9(3):471-9. doi: 10.1123/ijspp.2013-0390. Epub 2014 Feb 7. PMID 24509482
- [Background] Fatouros IG, Chatzinikolaou A, Douroudos II, Nikolaidis MG, Kyparos A, Margonis K, Michailidis Y, Vantarakis A, Taxildaris K, Katrabasas I, Mandalidis D, Kouretas D, Jamurtas AZ. Time-course of changes in oxidative stress and antioxidant status responses following a soccer game. J Strength Cond Res. 2010 Dec;24(12):3278-86. doi: 10.1519/JSC.0b013e3181b60444. PMID 19996787